CLINICAL TRIAL: NCT04565522
Title: Transmission of COVID-19 Among Patients and Health Personnel in Dialysis Centers: a Cohort Prospective Study (DIAL-COVID-19)
Brief Title: Transmission of COVID-19 Virus Among Patients and Staff in Dialysis Centers
Acronym: DIAL-COVID-19
Status: Completed | Type: Observational
Sponsor: Simeone Andrulli, MD (Other)
Responsible Party: Sponsor-Investigator, Simeone Andrulli, MD, Principal Investigator, A. Manzoni Hospital
Organization: A. Manzoni Hospital (Other)
Other Study IDs: DIAL-COVID-19
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Dialysis; Nurse-Patient Relations
Keywords: contact mapping
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hemodialysis or peritoneal dialysis patients: Hemodialysis or peritoneal dialysis Covid negative patients
  Interventions: Other: Prospective observation
- dialysis staff healthcare professionals: dialysis staff Covid negative healthcare professionals
  Interventions: Other: Prospective observation

INTERVENTIONS:
Other: Prospective observation — Prospective observation until one year follow-up

SUMMARY:
Patients on dialysis are at risk for several infectious diseases, since they have reduced immunological and have to regularly attend dialysis centres even if a pandemic is going on. Dialysis patients and healthcare professionals of dialysis centres can become infected one with the other. The incident risk of COVID-19 in dialysis centres is still unknown.

Given the challenges of an early diagnosis of COVID-19, the likely transmission with outbreaks, the possibility of reciprocal transmission of the infection among patients and healthcare professionals, the frequent clinical severity of COVID-19 in dialysis patients because of the coexistence of several comorbidities, CONTACT TRACING could be an effective and efficient tool to contrast COVID-19 spreading in dialysis centres.

DETAILED DESCRIPTION:
Patients on dialysis are at risk for several infectious diseases, since they have reduced immunological and have to regularly attend dialysis centres from once to thrice a week depending on their residual renal function even if a pandemic is going on.

Dialysis patients and healthcare professionals of dialysis centres can become infected one with the other.

The incident risk of COVID-19 in dialysis centres is still unknown. Given the challenges of an early diagnosis of COVID-19, the likely transmission with outbreaks, the possibility of reciprocal transmission of the infection among patients and healthcare professionals, the frequent clinical severity of COVID-19 in dialysis patients because of the coexistence of several comorbidities, CONTACT TRACING could be an effective and efficient tool to contrast COVID-19 spreading in dialysis centres. This modality keeps trace of the contacts the new COVID-19 case have had and allow the identification of other possible cases in that outbreak

Contact tracing is the key tool to detect and trace COVID-19 cases among patients and health care professionals, i.e. the space-time mapping of the contacts among these two categories:

1. Daily for healthcare professionals
2. At every dialysis session for haemodialysis patients
3. At every hospital visit for patients on peritoneal dialysis

Maximum follow will be up to 12 months excepting in those patients who develop a COVID-19-related clinically significant event:

1. Diagnosis of symptomatic COVID-19 with or without hospitalisation
2. Respiratory insufficiency with the need of CPAP or mechanical ventilation
3. Death associated or related to COVID-19

In the participating centres, the enrolment of patients and healthcare professionals will be prospective, progressive and competitive till the number of cases of COVD-19 will reach 200 subjects. If study participation will be 10% and COVID-19 will be taken by 4% of the patients with no prior exposure to COVID-19, we can estimate to enrol 5000 subjects (dialysis patients and healthcare professionals) over a period of 12 months in 50-150 centres. The length of the enrolment period of 6-12 months will depend also on future evolution of the pandemic in the Italian regions that have not been massively hit by the infection.

Study data will be stored on a web-database, which will be created on purpose. Privacy protection of patients and health care professionals will be pursued and granted by anonymous data collection.

Given the longitudinal and prospective design of the study, Kaplan-Meier curves will be used to describe the incidence of COVID-19 infection and the survival of dialysis patients and their healthcare professionals.

Cox multivariate analysis will be used to:

1. Estimate the incidence, morbidity and mortality of COVID-19 in the two categories
2. Estimate predictors and/or confounders associated with the incidence of the three study outcomes (infection, morbidity and mortality)

ELIGIBILITY:
Inclusion Criteria:

1. All the patients on haemodialysis or peritoneal dialysis giving their consent to participate
2. All healthcare professionals in charge of dialysis patients giving their consent to participate

Exclusion Criteria:

1. Dialysis patients or healthcare professionals who already have had Covid-19
2. Patients with kidney transplant
3. Patients with acute kidney injury (AKI) or on dialysis for less than 3 months
4. Life expectancy lower than 6 months
5. Patients already enrolled in other clinical trials
6. Absence of the consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients on haemodialysis
  2. Patients on peritoneal dialysis
  3. Healthcare professionals in charge of dialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 2847 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
incident risk of COVID-19 infection | 1 year
  incident risk of COVID-19 infection in dialysis patients and in related dialysis healthcare professionals

SECONDARY OUTCOMES:
Evaluate the morbidity of COVID-19 | 1 year
  Evaluate the morbidity (hospitalisation rate) of COVID-19 in the two subject categories
Evaluate the mortality of COVID-19 | 1 year
  Evaluate the mortality rate of COVID-19 in the two subject categories
Estimate the predictive role of comorbidities, inflammation indexes and therapy on the hospitalisation rate | Three months
  Estimate the predictive role of comorbidities, inflammation indexes and therapy on the hospitalisation rate in the three months after COVID-19 diagnosis
Estimate the predictive role of comorbidities, inflammation indexes and therapy on the mortality rate | Three months
  Estimate the predictive role of comorbidities, inflammation indexes and therapy on the mortality rate in the three months after COVID-19 diagnosis
Evaluate the infective role of dialysis staff towards patients | 1 year
  Evaluate the infective role of dialysis staff towards patients over one year follow-up
Evaluate the infective role of patients towards dialysis staff | 1 year
  Evaluate the infective role of patients towards dialysis staff over one year follow-up

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Cannizzaro, Catania
  - AOU Mater Domini, Catanzaro
  - AOU Careggi, Florence
  - Policlinico, Foggia
  - CEM-Mazara, Mazara del Vallo
  - Osp. San Francesco, Nuoro
  - SOS Nefrologia di Pescia, Pescia
  - Ospedale di Santo Stefano, Prato
  - Ambulatorio Dialisi di Tivoli, Roma
  - Geramed Srl, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Associazione Italiana Ricercare per Curare ODV ETS (AIRpC) — http://statgate.it